CLINICAL TRIAL: NCT02109913
Title: Phosphatidylinositol 3-kinase (PI3K) Pathway Analysis in Tumor Tissue and Circulating DNA to Obtain Further Insight in the Efficacy of Everolimus When Combined With Exemestane: A Side-study Protocol Attached to Standard Treatment With Everolimus and Exemestane for Postmenopausal Patients With Hormone Receptor-positive Advanced Metastatic Breast Cancer, Who Have Progressed on Anastrozole or Letrozole
Brief Title: Analysis of Tumor Tissue and Circulating Genetic Material in the Blood to Obtain Further Insight in the Effectiveness of Everolimus When Combined With Exemestane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Borstkanker Onderzoek Groep (Network); Novartis (Industry)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof dr Verheul, MD, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EudraCT 2013-004120-11; BOOG 2013-06 (Other: Dutch Breast Cancer Research Group (Borstkanker Onderzoek Groep; BOOG))
Record Dates: First submitted 2014-04-02; First posted 2014-04-10 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Hormone Receptor Positive Malignant Neoplasm of Breast; Metastatic Breast Cancer
Keywords: Breast Cancer; metastatic; hormone receptor positive; everolimus; biomarker
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus plus exemestane (Other): Biomarker study in patients receiving standard treatment
  Interventions: Drug: Everolimus plus Exemestane

INTERVENTIONS:
Drug: Everolimus plus Exemestane — Everolimus 10mg, oral, daily; exemestane 25 mg, oral, daily. Number of Cycles: until progression or unacceptable toxicity develops. From all patients, 4 additional blood samples, 6ml each, will be collected and an optional tumor biopsy will be taken, if eligible.
  Other Names: Afinitor; RAD001; CAS number 159351-69-6; EV Substance Code SUB02065MIG

SUMMARY:
The purpose of this study is to determine whether biomarkers could be found to gain more insight in tumor characteristics in order to predict which patients will have a high chance of a long progression-free survival. Postmenopausal patients with advanced metastatic breast cancer who have progressed on anastrozole or letrozole will be eligible for this study.

DETAILED DESCRIPTION:
Rationale of study:

Everolimus combined with exemestane has shown to improve progression-free survival compared to exemestane monotherapy in patients with hormone receptor-positive breast cancer previously treated with non-steroidal aromatase inhibitors. Since January 1st, 2013, everolimus is being reimbursed for this category of patients. For many patients this means, that an interesting treatment possibility has become available. However, some patients do not benefit from everolimus and exemestane, while others have to deal with side-effects requiring adjustment of the dose or even discontinuation of treatment.

In this study proposal the investigators plan to gain more insight in tumor characteristics in order to predict which patients will have a high chance of a long progression-free survival.

Study objectives:

1. It is proposed to compare progression-free survival on the combination of everolimus and exemestane between patients whose metastatic tumor expresses markers of phosphatidylinositol 3-kinase (PI3K) pathway activation versus patients whose metastatic tumor does not express PI3K pathway activation.
2. It is proposed to carry out immunohistochemistry on activated members of the PI3K pathway in primary tumor tissue of patients treated with everolimus and exemestane and compare the findings with the outcome of treatment and more specifically, with the results from other studies.
3. It is proposed to associate protein expression/ phosphorylation by proteomics in tumor biopsies to cancer mutations, PI3K pathway activation and progression-free survival on the exemestane and everolimus combination.
4. It is proposed to establish the incidence of mutations in phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) and protein kinase B (AKT) in peripheral blood of advanced breast cancer patients amenable for treatment with everolimus and exemestane and to explore whether the presence of such mutations is associated with outcome to treatment in these patients.

Study population:

Postmenopausal women with hormone receptor-positive locally advanced or metastatic breast cancer whose disease is refractory to non steroidal aromatase inhibitors (NSAIs) and have a documented recurrence or progression on last therapy for breast cancer.

Number of patients and centers:

* 175 patients for blood samples and archived tumor tissue, 50 for fresh tumor biopsy, another 30 for fresh tumor biopsy upon progressive disease
* 30 hospitals in the Netherlands.

Treatment phase:

Patients will be treated with 10 mg daily doses of everolimus (either 2 x 5 mg or 1 x 10 mg tablets) in combination with exemestane (25 mg daily tablets).

Dose adjustment (reduction, interruption) according to safety findings will be allowed.

Treatment will continue until one of the following conditions apply and whichever comes first: tumor progression, unacceptable toxicity according to investigator's judgment, patient's wish, death, discontinuation from the study for any other reason. Further treatment after progression will be at the investigator's discretion.

Physicians will collect data on demographics, previous treatments, efficacy of everolimus and exemestane as well as on toxic effects of this combination according to good clinical practice (GCP) in the patient's file.

Statistical considerations:

Since the majority of the studies involve the use of new techniques, the study will be mainly explorative in design. For blood sample analysis and analysis of archival tumor tissue at least 175 patients will be required. For tumor tissue biopsies a number of 50 patients is expected to give insight in differences between patients with clinical benefit ant those with early progressive disease; from 30 of these patients a tumor biopsy will be collected upon progressive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (≥ 18 years of age) with metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy.
2. Histological or cytological confirmation of estrogen-receptor positive (ER+) breast cancer
3. Postmenopausal women. Postmenopausal status is defined either by:

   * Age ≥ 55 years and one year or more of amenorrhea
   * Age < 55 years and one year or more of amenorrhea, with an estradiol assay < 40 pg/ml
   * Surgical menopause with bilateral oophorectomy
4. Disease refractory to NSAI, defined as:

   * a. Recurrence while on or within 12 months of end of adjuvant treatment with letrozole or anastrozole, or b. Progression while on or within one month of end of letrozole or anastrozole treatment for advanced breast cancer (locally advanced or metastatic )
   * Note: Letrozole or anastrozole do not have to be the last treatment prior to enrollment. Other prior anticancer therapy, e.g. tamoxifen, fulvestrant are allowed. Patients must have recovered to grade 1 or better from any adverse events (except alopecia) related to previous therapy prior to enrollment.
   * Radiological or clinical evidence of recurrence or progression on last systemic therapy prior to enrollment.
   * Note: There are no restrictions as to the last systemic therapy prior to enrollment.
5. Adequate bone marrow and coagulation function as shown by:

   * Absolute neutrophil count (ANC) ≥ 1.5 ×109/L
   * Platelets ≥ 100 ×109/L
   * Hemoglobin (Hgb) ≥ 5.6 mmol/L
   * INR (international normalized ratio) ≤ 2.0
6. Adequate liver function as shown by:

   * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN (upper limit of normal)(or ≤ 5 if hepatic metastases are present)
   * Total serum bilirubin ≤ 1.5 × ULN (≤ 3 × ULN for patients known to have Gilbert Syndrome)
7. Adequate renal function as shown by:

   - Serum creatinine ≤ 1.5 × ULN
8. Fasting serum cholesterol ≤ 7.75 mmol/L and fasting triglycerides ≤ 2.5 × ULN. In case one or both of these thresholds are exceeded, the patient can only be included after initiation of statin therapy or other lipid lowering drugs (eg fibrates), and when the above mentioned values have been achieved
9. Written informed consent obtained before any screening procedure and according to local guidelines.

Exclusion Criteria:

1. HER2-overexpressing patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive).
2. Previous treatment with mTOR (mammalian target of rapamycin) inhibitors.
3. Radiotherapy within four weeks prior to enrollment except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture which can then be completed within two weeks prior to enrollment. Patients must have recovered from radiotherapy toxicities prior to enrollment.
4. Currently receiving hormone replacement therapy, unless discontinued prior to enrollment.
5. Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use, at the time of study entry except in cases outlined below:
6. Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed.
7. Patients on stable low dose of corticosteroids for at least two weeks before enrollment are allowed in case of treatment of brain metastases.
8. Bilateral diffuse lymphangitic carcinomatosis or metastasis of the lung as the only manifestation of disease (>50% of lung involvement), evidence of metastases estimated as more than a third of the liver as defined by sonogram and/or CT scan.
9. Patients with a known history of HIV seropositivity.
10. Active, bleeding diathesis, or on oral anti-vitamin K medication (except low dose warfarin and acetylsalicylic acid or equivalent, as long as the INR is ≤ 2.0)
11. Any severe and / or uncontrolled medical conditions such as:

    * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to enrollment, serious uncontrolled cardiac arrhythmia
    * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 × ULN
    * Acute and chronic, active infectious disorders (except for hepatitis B and C positive patients) and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy
    * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
    * Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco (diffusing capacity of lung for carbon monoxide), O2 saturation at rest on room air should be considered to exclude restrictive pulmonary disease, pneumonitis or pulmonary infiltrates.
12. Patients who test positive for hepatitis B (HBV) or C (HBC) (patients who test negative for HBV-DNA, HBsAg, and HBcAb, but positive for HBsAb with prior history of vaccination against Hepatitis B will be eligible - see also 1.4)
13. Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (rifabutin, rifampicin, clarithromycin, ketoconazole, itraconazole, voriconazole, ritonavir, telithromycin) within the last 5 days prior to enrollment
14. History of non-compliance to medical regimens
15. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Biomarker Evaluation from Primary Tumor Tissue, New Tumor Biopsies and Blood Samples | Before start therapy until progression (expected average until progression: 11 months)
  Biomarker evaluation to gain more insight in tumor characteristics in order to predict which patients will have a high chance of a long progression-free survival. For biomarker evaluation, primary tumor tissue, new tumor tissue Biopsies and blood samples will be analysed for activated members of the PI3K pathway by immunohistochemistry and phosphoproteomics, and for the incidence of mutations in the PI3K pathway. The findings will be compared with the outcome of treatment and with the results from other studies.
Progression-free survival | From start therapy until first reported progression (expected average until progression: 11 months)
  Progression-free survival (PFS) is the time from date of start of treatment to the date of event defined as the first documented progression. Progressive disease will be assessed by radiological assessment or, if clearly stated in the patient's file, by clear clinical signs.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From start therapy until 28 days after progression (expected average until progression: 11 months)
  Adverse Events related to Everolimus will be recorded according to Common Toxicity Criteria for Adverse Effects (CTCAE) v4.03. Number of events and worst grades will be recorded, as well as reasons for dose reduction and discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Epie Boven, Prof.dr. MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (28):
- Netherlands (28):
  - VU University Medical Center, Amsterdam, North Holland
  - Flevoziekenhuis, Almere Stad
  - BovenIJ Ziekenhuis, Amsterdam
  - The Netherlands Cancer Institute, Amsterdam
  - Gelre, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Groep, Delft
  - Gemini, Den Helder
  - Deventer Ziekenhuis, Deventer
  - Maxima Medisch Centrum, Eindhoven
  - Groene Hart Ziekenhuis, Gouda
  - Tergooi ziekenhuizen, Hilversum
  - Spaarne Ziekenuis, Hoofddorp
  - MC Leeuwarden, Leeuwarden
  - LUMC, Leiden
  - Canisius Ziekenhuis, Nijmegen
  - Bravis, Roosendaal and Bergen Op Zoom
  - Erasmus University Medical Center, Rotterdam
  - Ikazia, Rotterdam
  - Vlietland, Schiedam
  - Orbis MC, Sittard
  - Haga, The Hague
  - MC Haaglanden, The Hague
  - Elisabeth - Tweesteden, Tilburg
  - UMC Utrecht, Utrecht
  - VieCuri, Venray
  - Isala, Zwolle

REFERENCES:
- [Background] Baselga J, Campone M, Piccart M, Burris HA 3rd, Rugo HS, Sahmoud T, Noguchi S, Gnant M, Pritchard KI, Lebrun F, Beck JT, Ito Y, Yardley D, Deleu I, Perez A, Bachelot T, Vittori L, Xu Z, Mukhopadhyay P, Lebwohl D, Hortobagyi GN. Everolimus in postmenopausal hormone-receptor-positive advanced breast cancer. N Engl J Med. 2012 Feb 9;366(6):520-9. doi: 10.1056/NEJMoa1109653. Epub 2011 Dec 7. PMID 22149876
- [Background] Yardley DA, Noguchi S, Pritchard KI, Burris HA 3rd, Baselga J, Gnant M, Hortobagyi GN, Campone M, Pistilli B, Piccart M, Melichar B, Petrakova K, Arena FP, Erdkamp F, Harb WA, Feng W, Cahana A, Taran T, Lebwohl D, Rugo HS. Everolimus plus exemestane in postmenopausal patients with HR(+) breast cancer: BOLERO-2 final progression-free survival analysis. Adv Ther. 2013 Oct;30(10):870-84. doi: 10.1007/s12325-013-0060-1. Epub 2013 Oct 25. PMID 24158787
- [Background] Lauring J, Park BH, Wolff AC. The phosphoinositide-3-kinase-Akt-mTOR pathway as a therapeutic target in breast cancer. J Natl Compr Canc Netw. 2013 Jun 1;11(6):670-8. doi: 10.6004/jnccn.2013.0086. PMID 23744866
- See also: EU Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-004120-11/NL
- See also: Dutch Breast Cancer Research Group (Borstkanker Onderzoek Groep; BOOG) — http://www.boogstudycenter.nl/home-15.html
- See also: VU University Medical Center — http://www.vumc.com/